CLINICAL TRIAL: NCT05070260
Title: A Randomized, Double Blind, Multicenter, Multinational, Placebo Controlled, Parallel Group, Single Dose, Adaptive Efficacy and Safety Study of Glenzocimab Used as an add-on Therapy on Top of Standard of Care un the 4.5 Hours Following an Acute Ischemic Stroke
Brief Title: ACTISAVE: ACuTe Ischemic Stroke Study Evaluating Glenzocimab Used as Add-on Therapy Versus placEbo
Acronym: ACTISAVE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Acticor Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ACT-CS-005
Record Dates: First submitted 2021-07-30; First posted 2021-10-07 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2023-08

CONDITIONS: Acute Ischemic Stroke
Keywords: Haemorrhages GPVI; Thrombolysis; Thrombectomy; Anti-platelet; glenzocimab; ACT017; stroke; GPVI
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — glenzocimab

STUDY DESIGN:
Intervention Model Description: A randomized, double blind, multicenter, multinational, placebo controlled, parallel group, single dose, adaptive phase II/III study (respectively Part 1 and 2).
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intravenous glenzocimab (ACT017) 1000 mg (Experimental): Intravenous glenzocimab (ACT017) 1000 mg to be added to thrombolysis +/- mechanical thrombectomy
  Interventions: Drug: Intravenous glenzocimab (ACT017) 1000 mg
- Intravenous Placebo (Placebo Comparator): Intravenous Placebo to be added to thrombolysis +/- mechanical thrombectomy
  Interventions: Drug: Intravenous Placebo

INTERVENTIONS:
Drug: Intravenous glenzocimab (ACT017) 1000 mg — Add-on therapy to the standard of Care in the treatment of the acute ischemic stroke symptoms
  Other Names: Thrombolysis +/- thrombectomy
  Arms: Intravenous glenzocimab (ACT017) 1000 mg
Drug: Intravenous Placebo — Add-on therapy to the standard of Care in the treatment of the acute ischemic stroke symptoms
  Other Names: Thrombolysis +/- thrombectomy
  Arms: Intravenous Placebo

SUMMARY:
A randomized, double blind, multicenter, multinational, placebo controlled, parallel group, single dose, adaptive phase II/III study.

The study evaluates the efficacy and safety of a fixed dose of glenzocimab (1000 mg IV over 6 hrs including initial bolus of 15 minutes) on top of the best standard of care.

DETAILED DESCRIPTION:
The study evaluates the efficacy and safety of a fixed dose of glenzocimab (1000 mg IV over 6 hrs including initial bolus of 15 minutes) on top of the best standard of care.

In all patients, the IVT should have been initiated prior to/at randomization, and in any case within 4.5 hrs post onset of acute ischemic stroke symptoms. IVT should mandatorily be used according to the approved dosing regimen as described in the product information/SmPC/USPI.

Eligible patients will be randomized and the infusion of glenzocimab or of its matching placebo should be administered as soon as possible but no later than two hours from the start of the thrombolytic agent administration. Transferring the patient to the catheterization room should not delay the Investigational Medicinal Product (IMP) administration.

Patients will be randomized in a 1:1 ratio allocation either to glenzocimab or placebo. Randomization will be minimized for factors as follows: (NIHSS <10 vs. ≥ 10), age group (<65, 65-79, ≥80 years), and type of thrombolytic agent (alteplase vs. tenecteplase) in order to balance each treatment group composition.

The allocation of each patient in all centers to an active treatment or placebo will strictly follow the central randomization scheme. Clinical supplies allocation to centers should provide the necessary material so that any eligible patient can receive the assigned treatment. A central randomization system (IRT - Interactive Response Technology) will be used to manage randomization/stratification and drug shipment. The whole process will be handled in a manner that it is blinded for the treatment received to all involved study personnel.

The IDMC will be composed of 5 independent members (at least 2 clinicians and 1 statistician).

IDMC members will process the information and will issue their recommendations as per the IDMC Charter.

One interim analysis after 100 patients recruited and treated is planned for safety evaluation only.

In case of any urgent safety concern, ad-hoc meetings will be triggered.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female patients ≥ 18 years (i.e., at least 18 years old at time of randomization)
2. Having given their own written consent, or legal representative consent, and in any case, in strict accordance with country-specific legal requirements,
3. Presenting with an acute disabling ischemic stroke either in the anterior or in posterior circulation, with or without visible occlusion, with a known time of onset, that is ≤ 4.5 hrs
4. Presenting with a pre-IVT NIHSS ≥ 6
5. In whom IVT is or has been initiated, whether or not patients are additionally eligible to mechanical thrombectomy (MT+ IVT), according to the recommendation of the last guidelines (ASA and ESO recommandations),
6. Women of childbearing potential (WOCBP) must have a negative serum/urine pregnancy test at baseline. Women of childbearing potential, i.e., fertile, are defined as women following menarche and until becoming post-menopausal unless permanently sterile, i.e., having undergone hysterectomy, bilateral salpingectomy and bilateral oophorectomy
7. Post-menopausal women defined as not having menses for 12 months without an alternative medical cause. For WOCBP, a highly effective birth control method should be in place that can achieve a failure rate of less than 1% per year that should last for at least 2 months after IMP administration.

   Birth control methods which may be considered as highly effective in WOCBP include:
   * combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (intravaginal, transdermal),
   * progestogen-only hormonal contraception associated with inhibition of ovulation (injectable, implantable)
   * intrauterine device (IUD),
   * intrauterine hormone-releasing system (IUS),
   * bilateral tubal occlusion,
   * vasectomized partner,

   Birth control methods which may be considered as highly effective for men and that should last for 4 months after IMP administration include:
   * vasectomy,
   * use of condom combined with a highly effective birth control method for their WOCBP partner.

   Please note that hormonal contraception is a risk factor for thromboembolic events and attention should be called to reconsider it passed the acute stroke phase.
8. Patients affiliated to a health insurance - modality depending on country legal requirement

Exclusion Criteria:

1. Coma, or NIHSS >25,
2. Patients < 18 years,
3. Protected adults under guardianship or curatorship,
4. Prior ischemic stroke within the past 3 months,
5. mRS pre-stroke known to be ≥ 2,
6. Large (more than 1/3 of the middle cerebral artery) regions of clear hypodensity on Baseline Computed Tomography Angiography (CTA) or Magnetic Resonance Imaging (MRI) or with vascular injection (MRA),
7. Significant mass effect with midline shift,
8. Stroke of hemorrhagic origin,
9. Patients likely to require dual antiplatelet therapy (DAPT) within the first 24 hrs after cessation of glenzocimab or placebo infusion for e.g., carotid stenting,
10. Known renal insufficiency (Grades 4-5 - severe or terminal with a creatinine clearance < 30 mL/min using Cockroft formula),
11. Known allergic reaction to contrast agents,
12. Patients under anti-coagulant therapy, except preventative doses of injectable low molecular weight heparin (LMWH),
13. Known ongoing treatment with a mAb,
14. Prior cardiopulmonary resuscitation < 10 days,
15. Childbirth within < 10 days,
16. Seizures at stroke onset if it precludes obtaining an accurate baseline (pre-IVT) NIHSS,
17. Life expectancy (except for stroke) < 3 months,
18. Pregnancy or breastfeeding,
19. Females of childbearing potential not using effective birth control methods,
20. Known current participation in another clinical investigation with experimental drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 438 (Actual)
Dates: Start 2021-09-23 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Binary Poor Outcome on the mRS defined by a score of 4-6 (versions 0-3) | Day 90
  To show the efficacy of glenzocimab vs. placebo, on the "poor outcome" defined as a mRS score of 4-6 (vs 0-3) assessed at Day 90

SECONDARY OUTCOMES:
Key Secondary Efficacy Endpoint - mRS | Day 90
  Binary "Favorable Outcome" on the mRS defined by a score of 0-2 (versus 3-6)
Mortality | Day 90
  All cause mortality
mRS | Day 90
  To assess the favorable responses defined as mRS score of 0-1
mRS | Day 90
  To assess the favorable responses defined as mRS score of 5-6
Ordinal mRS | Day 90
  To assess the shift analysis
Utility Weighted mRS | Day 90
  To assess the utility weighted mRS (UW-mRS)
All cause mortality | 72 hours
  To assess all cause mortality
ICHs | 72 hours
  Symptomatic and non-symptomatic ICHs
Neurological Status Change as assessed by NIHSS value compared to pre-IVT value | 24 hours
  Response defined by a relative decrease (%) in NIHSS value at 24 hours compared to pre-IVT value higher than 30%.
  Relative change (%) in NIHSS value at 24 hrs compared to pre-IVT value
Recanalization rate | Day 90
  To assess recanalization in patients undergoing thrombectomy by eTICI score
Cerebral tissue reperfusion | Day 90
  To assess Cerebral tissue reperfusion
Infarct volume progression and hemorrhagic transformation | 24 hrs
  To assess the impact on follow up imaging (follow up infarct volume, infarct growth and volume of hemorrhagic transformation)
Measure of Quality of Life by EuroQol-5 Dimension-5 Level (EQ-5D-5L) | Day 90
  Quality of Life as assessed by the EuroQol-5 Dimension-5 Level. A Quality-of-Life Scale (EQ-5D-5L)
Incidence of Deaths | Day 90
  Deaths within the first 24 hours and over the whole study period until Day 90 (Kaplan-Meier curve)
Incidence of Symptomatic intracranial hemorrhages | 24 hours
  Symptomatic intracranial hemorrhages, defined by both anatomical imaging (according to Heidelberg's classification) at the time of its occurrence associated with an increase in NIHSS score by 4 points or greater, or death that is not explained otherwise (according to ECASS III study definition (14))
Incidence of Non-symptomatic hemorrhages | 24 hours
  Non-symptomatic hemorrhages, seen on 24-hours plain CT-Scan, not present at baseline assessment, once other diagnoses are excluded
Incidence of Adverse Events, SAEs, bleeding-related events, and Treatment-Emergent Adverse Events (TEAEs) | Day 90
  Incidence, nature and severity of Adverse Events, SAEs, bleeding-related events, and Treatment-Emergent Adverse Events (TEAEs)
Change in vital signs (Blood Pressure) at any visit or discharge as compared to Baseline | 24 hours
  Blood Pressure will be assessed every 30 minutes during the 6 hours (infusion) then every 3 hours up to 24 hours.
Change in vital signs (Heart Rate) at any visit or discharge as compared to Baseline | 24 hours
  Heart Rate will be assessed every 30 minutes during the 6 hours (infusion) then every 3 hours up to 24 hours
Change in hematology assessments: RBC (Red Blood Cell Count) at 24 hours as compared to Baseline | 24 hours
  % of patient with change in RBC (Red Blood Cell Count) in million/mm3
Change in hematology assessments: RBC (Red Blood Cell Count) at Day 7 or discharge as compared to Baseline | Day 7
  % of patient with change in RBC (Red Blood Cell Count) in million/mm3
Change in hematology assessments: Hemoglobin at 24 hours as compared to Baseline | 24 hours
  % of patient with change in Hemoglobin in g/100ml
Change in hematology assessments: Hemoglobin at Day 7 or discharge as compared to Baseline | Day 7
  % of patient with change in Hemoglobin in g/100ml
Change in hematology assessments: Hematocrit at 24 hours as compared to Baseline | 24 hours
  % of patient with change in Hematocrit in %
Change in hematology assessments: Hematocrit at 24 hours at Day 7 or discharge as compared to Baseline | Day 7
  % of patient with change in Hematocrit in %
Change in hematology assessments: Mean Corpuscular Hemoglobin Volume (MCV) at 24 hours as compared to Baseline | 24 hours
  % of patient with change in Mean Corpuscular Hemoglobin Volume (MCV) in µ3
Change in hematology assessments: Mean Corpuscular Hemoglobin Volume (MCV) at Day 7 or discharge as compared to Baseline | Day 7
  % of patient with change in Mean Corpuscular Hemoglobin Volume (MCV) in µ3
Change in hematology assessments: Mean corpuscular hemoglobin content (MCHC) at 24 hours as compared to Baseline | 24 hours
  % of patient with change in Mean corpuscular hemoglobin content (MCHC) in pg
Change in hematology assessments: Mean corpuscular hemoglobin content (MCHC) at Day 7 or discharge as compared to Baseline | Day 7
  % of patient with change in Mean corpuscular hemoglobin content (MCHC) in pg
Change in hematology assessments: Corpuscular hemoglobin concentration (CHC) at 24 hours as compared to Baseline | 24 hours
  % of patient with change in Corpuscular hemoglobin concentration (CHC) in %
Change in hematology assessments: Corpuscular hemoglobin concentration (CHC) at Day 7 or discharge as compared to Baseline | Day 7
  % of patient with change in Corpuscular hemoglobin concentration (CHC) in %
Change in hematology assessments: Leucocytes(/mm3) at 24 hours as compared to Baseline | 24 hours
  % of patient with change in Leucocytes in /mm3
Change in hematology assessments: Leucocytes(/mm3) at Day 7 or discharge as compared to Baseline | Day 7
  % of patient with change in Leucocytes in /mm3
Change in hematology assessments: Platelets x 10^9 /L at 24 hours as compared to Baseline | 24 hours
  % of patient with change in Platelets x 10^9 /L
Change in hematology assessments: Platelets x 10^9 /L at 24 hours at Day 7 or discharge as compared to Baseline | Day 7
  % of patient with change in Platelets x 10^9 /L
Change biochemistry assessments : SGPT (Sérum Glutamate Pyruvate Transaminase) at 24 hours as compared to Baseline | 24 hours
  % of patient with change in SGPT in UI/L
Change biochemistry assessments : SGPT at Day 7 or discharge as compared to Baseline | Day 7
  % of patient with change in SGPT in UI/L
Change biochemistry assessments : SGOT at 24 hours as compared to Baseline | 24 hours
  % of patient with change in SGOT in UI/L
Change biochemistry assessments : SGOT at Day 7 or discharge as compared to Baseline | Day 7
  % of patient with change in SGOT in UI/L
Change biochemistry assessments: LDH at 24 hours as compared to Baseline | 24 hours
  % of patient with change in LDH in UI/l
Change biochemistry assessments : LDH at Day 7 or discharge as compared to Baseline | Day 7
  % of patient with change in LDH in UI/l
Change biochemistry assessments : Cholesterol at 24 hours as compared to Baseline | 24 hours
  % of patient with change in Cholesterol in g/L or mmol/L
Change biochemistry assessments : Cholesterol at Day 7 or discharge as compared to Baseline | Day 7
  % of patient with change in Cholesterol in g/L or mmol/L
Change biochemistry assessments : Triglycerid at 24 hours as compared to Baseline | 24 hours
  % of patient with change in Triglycerid in g/L or mmol/L
Change biochemistry assessments : Triglycerid at Day 7 or discharge as compared to Baseline | Day 7
  % of patient with change in Triglycerid in g/L or mmol/L
Change biochemistry assessments : Urea at 24 hours as compared to Baseline | 24 hours
  % of patient with change in Urea in g/L or mmol/L
Change biochemistry assessments : Urea at Day 7 or discharge as compared to Baseline | Day 7
  % of patient with change in Urea in g/L or mmol/L
Change biochemistry assessments : Creatinin at 24 hours as compared to Baseline | 24 hours
  % of patient with change in Creatinin in mg/L or µM/L
Change biochemistry assessments : Creatinin at Day 7 or discharge as compared to Baseline | Day 7
  % of patient with change in Creatinin in mg/L or µM/L
Change biochemistry assessments : GFR at 24 hours as compared to Baseline | 24 hours
  % of patient with change in GFR in mL/min/1,73 m²
Change biochemistry assessments : GFR at Day 7 or discharge as compared to Baseline | Day 7
  % of patient with change inGFR in mL/min/1,73 m²
Change biochemistry assessments : Serum Glucose at 24 hours as compared to Baseline | 24 hours
  % of patient with change in Serum Glucose in g/L
Change biochemistry assessments : Serum Glucose at Day 7 or discharge as compared to Baseline | Day 7
  % of patient with change in Serum Glucose in g/L
Change biochemistry assessments : D-Dimer at 24 hours as compared to Baseline | 24 hours
  % of patient with change in D-Dimer in µg/L
Change biochemistry assessments : D-Dimer at Day 7 or discharge as compared to Baseline | Day 7
  % of patient with change in D-Dimer in µg/L
Change biochemistry assessments : Fibrinogen at 24 hours as compared to Baseline | 24 hours
  % of patient with change in Fibrinogen in g/L
Change biochemistry assessments : Fibrinogen at Day 7 or discharge as compared to Baseline | Day 7
  % of patient with change in Fibrinogen in g/L
Change biochemistry assessments : INR score at 24 hours as compared to Baseline | 24 hours
  % of patient with change in INR Score
Change biochemistry assessments : INR score at Day 7 or discharge as compared to Baseline | Day 7
  % of patient with change in INR Score
Change biochemistry assessments : PT score at 24 hours as compared to Baseline | 24 hours
  % of patient with change in PT in sec
Change biochemistry assessments : PT score at Day 7 or discharge as compared to Baseline | Day 7
  % of patient with change in PT in sec
Change biochemistry assessments : aPTT score at 24 hours as compared to Baseline | 24 hours
  % of patient with change in aPTT in sec
Change biochemistry assessments : aPTT score at Day 7 or discharge as compared to Baseline | Day 7
  % of patient with change in aPTT in sec
Change in dipstick urinalysis assessments: Turbidity at 24 hours as compared to Baseline | 24 hours
  % of patient with change in Change in urinalysis assessments
Change in dipstick urinalysis assessments: pH at 24 hours as compared to Baseline | 24 hours
  % of patient with change in Change in urinalysis assessments
Change in dipstick urinalysis assessments: Glucose at 24 hours as compared to Baseline | 24 hours
  % of patient with change in Change in urinalysis assessments
Change in dipstick urinalysis assessments: Proteins at 24 hours as compared to Baseline | 24 hours
  % of patient with change in Change in urinalysis assessments
Change in dipstick urinalysis assessments: Blood at 24 hours as compared to Baseline | 24 hours
  % of patient with change in Change in urinalysis assessments
Change in dipstick urinalysis assessments: Leucocytes at 24 hours as compared to Baseline | 24 hours
  % of patient with change in Change in urinalysis assessments
Change in dipstick clinical laboratory assessments (urinalysis) at Day 7 or discharge as compared to Baseline | Day 7
  % of patient with change in Change in urinalysis assessments
Change in coagulation parameters (INR, PT, a PTT) | 24 hours
  Change in coagulation parameters (INR, PT, aPTT) at 24 hrs
ECG changes | 24 hours
  ECG change from baseline on QT, QTc, PR, ST and QRS intervals at 24 hours as compared to Baseline
ECG changes | Day 7
  ECG change from baseline on QT, QTc, PR, ST and QRS intervals at Day 7 as compared to Baseline
ECG changes | Day 90
  ECG change from baseline on QT, QTc, PR, ST and QRS intervals at discharge as compared to Baseline

OTHER OUTCOMES:
Imaging for exploratory endpoints | Baseline
  • Acute ischemic stroke diagnosis and occluded cerebral vessel identification assessed by CTA or MRA/MRI with Time of Flight (TOF) sequence at Baseline
Imaging for exploratory endpoints | 24 hours
  Non Symptomatic and Symptomatic intracranial hemorrhage detection assessed by a plain CT-scan or MRI at 24h

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Comenducci, MD, Study Director — Acticor Biotech
Locations (10):
- United States (9):
  - Black Medical center, Bradenton, Florida
  - Nova Clinical Research, Bradenton, Florida
  - Northside hospital, St. Petersburg, Florida
  - University of Chicago, Chicago, Illinois
  - Washington university, St Louis, Missouri
  - Miami Valley hospital, Dayton, Ohio
  - Chattanooga center for neurological research, Chattanooga, Tennessee
  - Houston Methodist hospital, Houston, Texas
  - Memorial Hermann Hospital, Houston, Texas
- University Clinic Essen, Essen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Voors-Pette C, Lebozec K, Dogterom P, Jullien L, Billiald P, Ferlan P, Renaud L, Favre-Bulle O, Avenard G, Machacek M, Pletan Y, Jandrot-Perrus M. Safety and Tolerability, Pharmacokinetics, and Pharmacodynamics of ACT017, an Antiplatelet GPVI (Glycoprotein VI) Fab. Arterioscler Thromb Vasc Biol. 2019 May;39(5):956-964. doi: 10.1161/ATVBAHA.118.312314. PMID 31017822
- [Background] Renaud L, Lebozec K, Voors-Pette C, Dogterom P, Billiald P, Jandrot Perrus M, Pletan Y, Machacek M. Population Pharmacokinetic/Pharmacodynamic Modeling of Glenzocimab (ACT017) a Glycoprotein VI Inhibitor of Collagen-Induced Platelet Aggregation. J Clin Pharmacol. 2020 Sep;60(9):1198-1208. doi: 10.1002/jcph.1616. Epub 2020 Jun 4. PMID 32500636
- [Derived] Pottecher J, Raffi F, Jandrot-Perrus M, Binay S, Comenducci A, Desort-Henin V, Francois D, Gharakhanian S, Labart M, Meilhoc A, Toledano E, Pletan Y, Avenard G, Sato VH; GARDEN Investigators. Targeting GPVI with glenzocimab in COVID-19 patients: Results from a randomized clinical trial. PLoS One. 2024 Jun 17;19(6):e0302897. doi: 10.1371/journal.pone.0302897. eCollection 2024. PMID 38885234